CLINICAL TRIAL: NCT06349564
Title: Pilot Proof of Concept Study for Implementing Virtual Reality (VR) to Reduce Sedation Requirement During Endoscopy
Brief Title: Implementing Virtual Reality (VR) to Reduce Sedation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-01443
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Sedative During Endoscopy
Keywords: GERD; Dyspepsia; screening colonoscopy; diagnostic upper endoscopy; Gastroesophageal reflux disease
MeSH Terms: conditions — Gastroesophageal Reflux; Dyspepsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic Procedure with VR Headset (Experimental): VR google with noise cancellation headphones will be placed on patients' heads after a time-out. Patients can select from a range of entertainment videos prior and during the procedure. The anesthesiologist will administer minimal sedation. The patient can request additional sedation if needed. VR immersion continues until the procedure concludes and patients are moved to the recovery area. Goggles are removed in the recovery area
  Interventions: Device: Pico 4 Enterprise headset with noise cancelling headphones
- Endoscopic Procedure only (No Intervention): The control group will be chart review of patients undergoing similar endoscopic procedure from November 30, 2023 to June 31st, 2023.

INTERVENTIONS:
Device: Pico 4 Enterprise headset with noise cancelling headphones — The device includes a computer tablet and virtual reality headset.
  Arms: Endoscopic Procedure with VR Headset

SUMMARY:
The study is a prospective pilot patients aged 21 to 65 undergoing screening colonoscopy or diagnostic upper endoscopy. Patients are administered minimal sedation (2 mg of Versed and 25 mg of Fentanyl) and are given Virtual Reality (VR) goggles to wear for the duration of the procedure. The purpose of this study is to assess the feasibility, effect, and safety of using VR goggles during endoscopic procedures to decrease sedation requirements, enhance patient satisfaction, and reduce recovery time.

ELIGIBILITY:
INTERVENTION GROUP

Inclusion Criteria:

* Undergoing screening colonoscopy or diagnostic upper endoscopy for GERD or dyspepsia at NYU Langone Brooklyn Hospital
* Aged 21 to 65

Exclusion Criteria:

* Visual impairments such as blindness which would impair them from watching the entertainment videos.
* Patients with history of CAD,
* History of seizures,
* History of vertigo,
* History of allergy to plastic,
* ASAII or III,
* Patient with active GI bleed, having either melena or hematochezia.

CONTROL GROUP

Inclusion Criteria:

* Underwent screening colonoscopy or diagnostic upper endoscopy for GERD or dyspepsia at NYU Langone Brooklyn Hospital
* Aged 21 to 65

Exclusion Criteria:

* Visual impairments such as blindness which would impair them from watching the entertainment videos
* Patients with history of CAD
* History of seizures
* History of vertigo
* History of allergy to plastic
* ASAII or III
* Patient with active GI bleed, having either melena or hematochezia

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Total amount of sedative drugs administered during the procedure | End of procedure, up to 1 hour

SECONDARY OUTCOMES:
Patient-reported discomfort or pain (using 0-10 pain scale) | During PACU stay, approximately 30 minutes
Duration of the procedure | End of procedure, up to 1 hour
Overall patient satisfaction scores | During PACU stay, approximately 30 minutes
  Using Likert scale of 1-7. Subjects will be asked to rank several variables on the Likert scale, including overall experience (from 1-very dissatisfied to 7-very satisfied), enjoyability (from 1- not enjoyable to 7-very enjoyable), and anxiety (from 1-extreme anxiety to 7-no anxiety). Scores range from 3-21, higher scores indicate satisfaction.
Number of events of complications from VR | During PACU stay, approximately 30 minutes
  Events such as nausea, vomiting, dizziness.
Number of technical failures | End of procedure, up to 1 hour
Troubleshooting time | End of procedure, up to 1 hour
PACU length of stay | End of PACU stay, approximately 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Maysaa El Zoghbi, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Brooklyn, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Maysaa.ElZoghbi@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to Maysaa.ElZoghbi@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.